CLINICAL TRIAL: NCT05833737
Title: Corneal Findings in Patients Treated With Belantamab Mafodotin - a Prospective Study Focusing on Corneal Nerves
Brief Title: Corneal Findings in Patients Treated With Belantamab Mafodotin
Status: Terminated | Type: Observational
Why Stopped: Study medication market withdrawal by FDA.
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julia Aschauer, Principal Investigator, Medical University of Vienna
Other Study IDs: CoFiBe2023
Record Dates: First submitted 2023-04-11; First posted 2023-04-27 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma; Corneal Diseases; Corneal Cyst
MeSH Terms: conditions — Multiple Myeloma; Corneal Diseases | interventions — belantamab mafodotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Belantamab mafodotin — Injection for refractory/relapsed multiple myeloma

SUMMARY:
In the upcoming years, more and more ophthalmologists will be confronted with patients receiving Belantamab mafodotin (Belamaf) treatment due to the promising effects on survival in multiple myeloma patients. Early, at best subclinical detection of corneal damage may contribute to the definition of the optimal dosing regimen as well as therapy interval in each patient without the need to stop this lifesaving treatment. However, until today, studies focusing on the development, morphology, and evolution of corneal epithelial changes associated with Belamaf treatment are scarce. In order to clarify the precise pathomechanism of the associated keratopathy, innovative imaging techniques such as corneal confocal microscopy (CCM) need to be used to follow patients prior to therapy and on a regular basis during treatment intervals. In specific, different regions of the cornea, including the central apex, the (mid-) periphery and the limbus need to be explored. The latter, in specific, is often claimed to play an important role in the uptake of Belamaf into the cornea, but has not been studied in any approach so far.

Likewise, there are no reports on the effects of Belamaf on corneal layers adjacent to the corneal epithelium, in specific the subepithelial nerve plexus (SNP). Changes in this layer may suggest a potential peripheral neurotoxic/neurodegenerative effect, associated with Belamaf.

Furthermore, there is a lack of evidence from literature on how changes in the anterior layers of the cornea as studied with confocal microscopy in patients on Belamaf treatment differ from distinct corneal changes in these same layers in patients with other anterior corneal diseases including keratokonjunctivits sicca, epithelium basement membrane dystrophy and limbal stem cell disease.

At last, regeneration of the corneal surface after Belamaf discontinuation has been described and is expected, but detailed information on the time to corneal rehabilitation as well as confocal microscopic follow-up of epithelial and neuronal layers during this time is warranted. The purpose of this monocentric, prospective longitudinal study is to answer these specific research questions in a combined clinical approach using corneal confocal microscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
2. Participant must be ≥ 18 years of age at the start of belantamab mafodotin treatment
3. Confirmed diagnosis of multiple myeloma
4. Due to receive belantamab mafodotin per routine clinical care by a hematologist consistent with the approved labelling (received at least four prior therapies and whose disease is refractory to at least one proteasome inhibitor, one immunomodulatory agent, and an anti-CD38 monoclonal antibody, and who have demonstrated disease progression on the last therapy). The inclusion will be based on the clinical judgement of the hematologists and the estimation about the patient´s ability to co-operate during the ophthalmological examinations. All inclusion and exclusion criteria for belamaf medication are upon judgment of the prescribing hematooncologist and are therefore not part of this study protocol.

Exclusion Criteria:

1. Participant must not have any signs of corneal disease before study entry.
2. As stated above, the inclusion and exclusion criteria for belamaf medication are upon judgment of the prescribing hemato-oncologist, and are therefore not part of this study protocol.
3. Uncontrolled glaucoma
4. Medical history of (diabetic) polyneuropathy
5. Inability to comply with follow-up visits
6. Participant must not have known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include about 50 consecutive patients referred from the Department of Internal Medicine I, Division of Hematology and Hemostaseology, who are scheduled for treatment with Belamaf due to multiple myeloma. Patients will be receiving Belamaf per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
change in corneal nerve fibre density (CNFD) treatment using | three weeks after completion of the third cycle of Belamaf infusion
  change in CNFD measured with confocal microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No